CLINICAL TRIAL: NCT06873022
Title: Electromyography Biofeedback and Neuromuscular Electrical Stimulation of Deltoid in Patients With Reverse Total Shoulder Arthroplasty
Brief Title: EMG Biofeedback and NMES of Deltoid in Patients With rTSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 202403141DINE
Record Dates: First submitted 2025-02-17; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2024-05

CONDITIONS: Reverse Shoulder Replacement
Keywords: reverse total shoulder arthroplasty; neuromuscular electrical stimulation; surface electromyography; biofeedback; scapulohumeral rhythm
MeSH Terms: interventions — Biofeedback, Psychology

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- biofeedback (Experimental): sEMG biofeedback: Subjects were instructed to monitor the sEMG signals of the D/UT balances ratio on the screen and maintain the D/UT balances ratio above the threshold during arm elevation and lowering. The threshold was set at 1 standard deviation of the ratio average at baseline (before intervention).
  Interventions: Device: biofeedback
- neuromuscular electrical stimulation (Experimental): NMES: Two electrode pads were placed on the anterior, middle, and posterior deltoid boundary lines and at a distance of 1cm distal to the lateral margin of the acromion. The operator palpated the deltoid muscle contraction and asked the subjects to perform arm elevation task with NMES. (frequency of 35 Hz and a duration of 250 microseconds.) A verbal cue was given during both th A verbal cue was given during both the sEMG biofeedback and NMES interventions: "Lengthen your arm as if you want to touch the ground, the scapula keeps in the neutral position, and then elevate your arm." Each intervention consisted of 3 sets of 10 repetitions per set, with a 1-minute rest between sets.
  Interventions: Device: neuromuscular electrical stimulation

INTERVENTIONS:
Device: neuromuscular electrical stimulation — NMES: Two electrode pads were placed on the anterior, middle, and posterior deltoid boundary lines and at a distance of 1cm distal to the lateral margin of the acromion. The operator palpated the deltoid muscle contraction and asked the subjects to perform arm elevation task with NMES. (frequency of 35 Hz and a duration of 250 microseconds.) A verbal cue was given during both th
  A verbal cue was given during both the sEMG biofeedback and NMES interventions: "Lengthen your arm as if you want to touch the ground, the scapula keeps in the neutral position, and then elevate your arm." Each intervention consisted of 3 sets of 10 repetitions per set, with a 1-minute rest between sets.
  Arms: neuromuscular electrical stimulation
Device: biofeedback — sEMG biofeedback: Subjects were instructed to monitor the sEMG signals of the D/UT balances ratio on the screen and maintain the D/UT balances ratio above the threshold during arm elevation and lowering. The threshold was set at 1 standard deviation of the ratio average at baseline (before intervention).
  Arms: biofeedback

SUMMARY:
The effect of NMES and surface electromyography (sEMG) biofeedback on the deltoid and associated scapular muscles in scapular kinematics and muscle activation in individual post rTSA

DETAILED DESCRIPTION:
Reverse total shoulder arthroplasty (rTSA) has been the optimal treatment for massive irreparable rotator cuff tears and cuff tear arthropathy. Since scapular kinematics alteration was associated with shoulder disorders, scapular kinematics had been characterized in individuals post rTSA with more upward rotation, external rotation, and posterior tilt of the scapula. In addition, the average scapulohumeral rhythm ranged from 1.1 to 1.6, indicating lower glenohumeral joint movements and higher scapulothoracic movements. It supposed that more scapula upward rotation without adequate humeral elevation can result in the scapula notching. Therefore, strategy to decrease scapular movement or increase humeral movements during arm movements may prevent scapula notching. To compensate for rotator cuff deficiency, the deltoid muscle plays a crucial role post rTSA. Enhancing deltoid function can be accomplished through the use of biofeedback or neuromuscular electrical stimulation (NMES). However, the effect of NMES and surface electromyography (sEMG) biofeedback on the deltoid and associated scapular muscles in scapular kinematics, muscle activation, and muscle balance ratio in individual post rTSA remained unclear. Therefore, the objectives in this study would to (1) determine the immediate effects of NMES with EMG biofeedback to deltoid (D) on the muscle activation of upper trapezius (UT), lower Trapezius (LT) and serratus Anterior (SA) as well as the scapular kinematics (upward/downward rotation, external/internal rotation, anterior/posterior tilting) (2) evaluate the immediate effects of NMES with EMG biofeedback on the muscle balance ratios (D/UT, D/LT, D/SA) and the scapulohumeral rhythm (SHR) during arm elevation in the scapular plane at different range of motion.

ELIGIBILITY:
Inclusion Criteria:

* (1) age between 20 to 85 years old
* (2) undergoing primary reverse shoulder arthroplasty
* (3) shoulder abduction in scapular plane above 90 degrees
* (4) above 3 months following rTSA

Exclusion Criteria:

* (1) a history of other shoulder surgery on the rTSA shoulder
* (2) a revision rTSA
* (3) a surgery shoulder muscle tendon transfer
* (4) neuromuscular diseases
* (5) cognitive disorders
* (6) contraindications for NMES

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2025-05-20 (Estimated); Study Completion 2025-05-20 (Estimated)

PRIMARY OUTCOMES:
Muscle activation | before intervention (baseline) and through intervention completion, an average 15 minutes in each intervention (sEMG biofeedback or NMES)
  Muscle activation The muscle activation of upper trapezius, lower trapezius, serrates anterior, and deltoid were collected during arm elevation task by sEMG at baseline, post- sEMG biofeedback, and post- NMES. Muscle activation was analyzed based on 0°-30°, 30°-60°, and 60°-90° during arm elevation and lowering. The sEMG data was calculated using the root mean square (RMS) based on average of middle three from five trials. The MVIC of UT, LT, SA, and D were used to normalize the sEMG data.
Scapular kinematics | before intervention (baseline) and through intervention completion, an average 15 minutes in each intervention (sEMG biofeedback or NMES)
  Scapular kinematics The scapular kinematics during arm elevation task was captured using an electromagnetic motion analysis system. The three scapula orientations were described using the Euler angle sequence with an X-axis for scapular posterior/anterior tilt, Y-axis for scapular upward/downward rotation, and Z-axis for scapular internal/external rotation. The average of middle three from five trials on scapular kinematics were analyzed at 30°, 60°, and 90° arm elevation and lowering.

SECONDARY OUTCOMES:
Muscle balance ratios | before intervention (baseline) and through intervention completion, an average 15 minutes in each intervention (sEMG biofeedback or NMES)
  Muscle balance ratios The muscle balance ratios of D/UT, D/LT, and D/SA were calculated based on average of middle three from five trials at the phases of 0°-30°, 30°-60°, and 60°-90° during arm elevation and lowering phase.
Scapulohumeral rhythm | before intervention (baseline) and through intervention completion, an average 15 minutes in each intervention (sEMG biofeedback or NMES)
  Scapulohumeral rhythm The scapulohumeral rhythm data was collected by humeral elevation relative to scapular upward rotation at the phases of 30°, 60°, and 90° arm elevation and lowering in scapular plane. The data was based on average of middle three from five trials.

CONTACTS AND LOCATIONS:
Overall Officials: Jiu-Jenq Lin, Ph.D, Study Chair — School and Graduate Institute of Physical Therapy, College of Medicine, National Taiwan University, Taipei, Taiwan
Locations (1):
- National Taiwan University of school and graduate of physical therapy of Performance Analysis Laboratory, Taipei, Zhongzheng Dist., Taiwan

IPD SHARING:
Plan to Share IPD: No